CLINICAL TRIAL: NCT04879537
Title: Optimized Acute Care for Geriatric Patients Using an Intersectoral Telemedical Cooperation Network - Around the Clock
Acronym: Optimal@NRW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Optimal@NRW Research Group (Unknown)
Responsible Party: Principal Investigator, Jörg Christian Brokmann, PD Dr. med., RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 19-019
Record Dates: First submitted 2021-03-31; First posted 2021-05-10 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Emergencies
Keywords: telemedicine; geriatric; early warning score; acute care; nursing home; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: Stepped-Wedge-Design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in this group are routinely treated.
- Telemedical support (Active Comparator): Participants in this group are routinely treated with additional telemedical support and the use of the early warning system.
  Interventions: Other: Telemedical support

INTERVENTIONS:
Other: Telemedical support — The nursing homes participating in the project will be equipped with telemedical equipment. This will allow teleconsultations to take place when needed. In addition, an early warning system will be introduced and, within the framework of the teleconsultation, a trained medical assistant can be sent to the care facility if necessary, who can carry out medical activities on site under a physician's delegated instructions. In addition, an electronic patient file will be introduced which can be accessed by the telemedicine physician and the general practitioner.
  Arms: Telemedical support

SUMMARY:
Due to "demographic change", the composition of the population in Germany is changing. The consequence of this change is a population that is getting older on average. A key challenge is the appropriate nursing and medical care of older people in senior residences and care facilities. The increasing workload for nursing staff and doctors in the outpatient sector means that timely care for patients, e.g. in the form of GP visits, cannot always be guaranteed in a timely manner. The results are unnecessary or premature hospital admissions as well as ambulance and emergency care interventions, even though in many cases it is not an acute or even life-threatening event. Furthermore, it has been scientifically proven that hospital admissions can increase the risk of patients becoming confused. The aim of this project is to avoid unnecessary hospital admissions and to enable patients to remain in their familiar surroundings as far as this appears medically justifiable. At the same time, the study aims to improve the medical care of nursing home residents through better networking of medical areas, the use of tele-consultations and an early warning system.

DETAILED DESCRIPTION:
The Optimal@NRW project represents a new cross-sectoral approach to the acute care and support of geriatric people in need of care through the implementation of an early warning system and the integration of a telemedical consultation system in 25 nursing homes in the region of Aachen in Germany. The project focuses on restructuring emergency care in nursing homes and improving cooperation between the actors involved (emergency service, emergency department, general practitioners, nursing staff, etc.). Accordingly, a central emergency number of the statutory health insurance funds is to act as a virtual hub for the care of geriatric patients.

The concrete approach of the project is that the participating nursing homes first contact the medical call centre (116 117) in case of a medical problem. The call centre is then responsible for an initial medical assessment and decides whether the respective GP can be called in or whether a teleconsultation with the "virtual digital desk" (i.e. the medical experts from the emergency department of the University Hospital RWTH Aachen) should be carried out. In addition, mobile nursing assistants (NÄPÄ (Z)) will be introduced as part of the project, who can also support the nursing staff and provide services that can be delegated by doctors - especially if the general practitioner is not available at the time.

In addition, a standardised early warning system is to be established in the nursing homes and its benefits evaluated. This will enable potentially dangerous changes in the state of health of nursing home residents to be detected earlier.

ELIGIBILITY:
Inclusion Criteria:

* Resident of one of the participating nursing homes
* At least 18 years old
* Written informed consent
* Consent of the guardian for residents who are not legally able to give consent

Exclusion Criteria:

* Persons placed in an institution by order of an authority or court
* Persons who are in a dependent or employment relationship with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Days spent at hospital | 24 months
  Days spent at hospital
Number of Intervention-related adverse events | 6 to 15 months depending on the cluster affiliation
  * Resuscitation during teleconsultation
  * Unexpected death during teleconsultation
  * Unexpected death within 24 hours after teleconsultation
  * Unexpected hospitalisation within 24 hours of teleconsultation
  * Unexpected death while wearing a biosensor (if available)

SECONDARY OUTCOMES:
Days spent at nursing home | 24 months
  Days spent at nursing home
Number of medical contacts | 24 months
  Number of medical contacts
Time to doctor contact | 24 months
  Time to doctor contact
Number of admissions to hospital | 24 months
  Admission to hospital in general and to specific diagnosis
Amount of use of medical services | 24 months
  Use of medical services
Number of ambulatory sensitive hospital cases | 24 months
  Number of ambulatory sensitive hospital cases
Cost effects via HCRU | 24 months
  Cost effects via HCRU
Transport units used | 24 months
  Transport units used
Quality of Life - QOL-AD | 24 months
  Quality of life assessed using Quality of Life-Alzheimer's Disease (QoL-AD). The total score ranges from 13 to 52, with a higher number indicating better quality of life
Quality of Life - VR-12 | 24 months
  Quality of life assessed using Veterans Rand 12 Item Health Survey (VR-12). The outcome includes a physical and mental health component score (PCS and MCS, respectively). Each component score (PCS and MCS) has a range of 0-100, with a higher score on the PCS and MCS indicating better outcome, or better physical or mental health-related quality of life, respectively.
Barthel Index | 24 months
  Assessment procedures of daily living skills assessed via Barthel Index. Score of the Barthel Index ranging from 0 to 100 were collected when 0 is the minimum (worst outcome) and 100 is the maximum (best outcome).
Dementia Screening Scale (DSS) | 24 months
  Identification of people with dementia syndromes in inpatient care for the elderly using Dementia Screening Scale (DSS). Score of the DSS ranging from 0 to 14. When 0 is the minimum (no impairment) and 14 is the maximum (maximum impairment).
Number of double prescriptions | 24 months
  Number of double prescriptions (drug therapy safety)
Number of hospitalizations due to medication | 24 months
  Number of hospitalizations due to medication (drug therapy safety)
Number of adverse events due to medication | 24 months
  Number of adverse events due to medication (drug therapy safety)
Time-to-event concerning medication and hospitalization | 24 months
  Time-to-event concerning medication and hospitalization (drug therapy safety)
Need for additional staff in case of telemedical call | 24 months
  Need for additional staff in case of telemedical call
Amount of ambulance service calls | 24 months
  Amount of ambulance service calls
hospital referrals and use of primary care physicians and physicians of the GP emergency service before and after the implementation of telemedicine in nursing homes | 9 to 18 months depending on the cluster affiliation
  hospital referrals and use of primary care physicians and physicians of the GP emergency service before and after the implementation of telemedicine in nursing homes
Response times in doctor-patient contact | 24 months
  Response times in doctor-patient contact before and after the implementation of telemedicine in nursing homes
Number of incorrect suspected diagnoses compared to diagnoses after teleconsultation or admission to hospital | 24 months
  - Number of most diagnosed diseases with correct/incorrect suspected diagnoses
Number of incorrect suspected diagnoses compared to diagnoses after teleconsultation or admission to hospital | 24 months
  - Concordance rate of suspected and confirmed diagnoses related to specific diseases
Number of incorrect suspected diagnoses compared to diagnoses after teleconsultation or admission to hospital | 24 months
  - Causes of inaccurate suspected diagnoses
Rate of guideline deviations in diagnostics and therapy for specific tracer diagnoses (e.g. hypertension/blood pressure derailment, blood sugar derailment, infections - community-acquired (urinary tract infection, bronchitis, pneumonia)) | 24 months
  Reasons for deviations (lack of knowledge, individual knowledge about patient, allergies, living will, local conditions/treatment resources, patient wishes)
Evaluation of the processes, NÄPA (Z) operations and tele consultations | 6 to 15 months depending on the cluster affiliation
  - Number of operations
Evaluation of the processes, NÄPA (Z) operations and tele consultations | 6 to 15 months depending on the cluster affiliation
  - Number of a new teleconsultation during or after a NÄPÄ (Z) operation
Evaluation of the processes, NÄPA (Z) operations and tele consultations | 6 to 15 months depending on the cluster affiliation
  - Need for hospitalization
Evaluation of the processes, NÄPA (Z) operations and tele consultations | 6 to 15 months depending on the cluster affiliation
  - Misadmissions
Evaluation of the processes, NÄPA (Z) operations and tele consultations | 6 to 15 months depending on the cluster affiliation
  Number of deviations between initially defined catalogue of requirements and acutal requirements
Evaluation of the processes, NÄPA (Z) operations and tele consultations | 6 to 15 months depending on the cluster affiliation
  - Point of time of the operations
Evaluation of the processes, NÄPA (Z) operations and tele consultations | 6 to 15 months depending on the cluster affiliation
  - Duration of the operations
Evaluation of the processes, NÄPA (Z) operations and tele consultations | 6 to 15 months depending on the cluster affiliation
  - Number of request by primary care physician, primary care emergency service, tele physician
Evaluation of the processes, NÄPA (Z) operations and tele consultations | 6 to 15 months depending on the cluster affiliation
  Questionnaire about the acceptance of nursing home staff
Applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  - Number of false alarms
Applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  - Number of measurements with the spot-check monitor
Applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  - rate of accuracy in detecting a deterioration in health condition
Applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  - Rate of different parameters leading to an diagnosis
Applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  - frequency of diagnosis derived from the early warning system
Applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  Questionnaire or interview to survey acceptance by caregivers and residents
Applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  Questionnaire or interview to survey the usability
Applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  Incidence of parameters leading to alarm/decisive parameters
Applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  Incidence of correct recognition of deteriorating medical conditions
Rate of applicability of an early warning score in nursing homes | 6 to 15 months depending on the cluster affiliation
  - tracer-diagnoses: fever, urinary-tract infection, pneumonia, cardiac decompensation, cardiac arrhythmia, reduced vigilance, hypertension, hypo-/hyperglycaemia, pain
Gender differences | 24 months
  Gender differences

OTHER OUTCOMES:
Satisfaction survey | 24 months
  Questionnaires to survey satisfaction about the intervention in the project
Satisfaction survey | 24 months
  Interviews to survey satisfaction about the intervention in the project
Ethic survey | 24 months
  Questionnaires to clarify whether the intervention is seen as ethically appropriate
Ethic survey | 24 months
  Interviews to clarify whether the intervention is seen as ethically appropriate
Acceptance survey | 24 months
  Questionnaires to survey acceptance about the intervention in the project
Acceptance survey | 24 months
  Interviews to survey acceptance about the intervention in the project

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Christian Brokmann, PD Dr. med., Principal Investigator — Uniklinik RWTH Aachen
Locations (1):
- University Hospital RWTH Aachen, Aachen, Germany

REFERENCES:
- [Background] Brown CA, Lilford RJ. The stepped wedge trial design: a systematic review. BMC Med Res Methodol. 2006 Nov 8;6:54. doi: 10.1186/1471-2288-6-54. PMID 17092344
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] Hoffmann F, Schmiemann G. Influence of age and sex on hospitalization of nursing home residents: A cross-sectional study from Germany. BMC Health Serv Res. 2017 Jan 19;17(1):55. doi: 10.1186/s12913-017-2008-7. PMID 28103927
- [Background] Sundmacher L, Fischbach D, Schuettig W, Naumann C, Augustin U, Faisst C. Which hospitalisations are ambulatory care-sensitive, to what degree, and how could the rates be reduced? Results of a group consensus study in Germany. Health Policy. 2015 Nov;119(11):1415-23. doi: 10.1016/j.healthpol.2015.08.007. Epub 2015 Sep 2. PMID 26428441
- [Background] Vossius C, Selbaek G, Saltyte Benth J, Bergh S. Mortality in nursing home residents: A longitudinal study over three years. PLoS One. 2018 Sep 18;13(9):e0203480. doi: 10.1371/journal.pone.0203480. eCollection 2018. PMID 30226850
- [Background] Bundesärztekammer. Beschlussprotokoll des 121. Deutschen Ärztetages in Erfurt vom 08. bis 11.05.2018, Stand 08.06.2018.
- [Background] Eatock D. Demografischer Ausblick für die Europäische Union 2019.
- [Background] Fehr A, Lange C, Fuchs J, Neuhauser H, Schmitz R. Gesundheitsmonitoring und Gesundheitsindikatoren in Europa. Robert Koch-Institut, Epidemiologie und Gesundheitsberichterstattung; 2017.
- [Background] Jacobs K, Kuhlmey A, Greß S, Klauber J, Schwinger A. Pflege-Report 2018. Berlin, Heidelberg: Springer Berlin Heidelberg; 2018.
- [Background] Sachverständigenrat zur Begutachtung der Entwicklung im Gesundheitswesen. Bedarfsgerechte Steuerung der Gesundheitsversorgung. Gutachten 2018.
- [Derived] Brucken D, Unterkofler J, Pauge S, Bienzeisler J, Hubel C, Zechbauer S, Rossaint R, Greiner W, Aufenberg B, Rohrig R, Bollheimer LC; Optimal@NRW Research Group; Brokmann JC. Optimal@NRW: optimized acute care of nursing home residents using an intersectoral telemedical cooperation network - study protocol for a stepped-wedge trial. Trials. 2022 Sep 27;23(1):814. doi: 10.1186/s13063-022-06613-1. PMID 36167557